CLINICAL TRIAL: NCT03488654
Title: The Heart in Systemic Lupus Erythematosus - a Comprehensive Approach by Cardiovascular Magnetic Resonance Tomography
Brief Title: CMR-Lupus Comprehensive Approach by Cardiovascular Magnetic Resonance Tomography
Status: Terminated | Type: Observational
Why Stopped: Recruitement problems as single centre study
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Heart-SLE
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Lupus Erythematosus, Systemic; Coronary Artery Disease; Myocardial Disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Coronary Artery Disease; Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance — CMR including cine, late gadolinium enhancement (LGE) and stress perfusion sequences

SUMMARY:
In systemic lupus erythematosus (SLE), cardiac manifestations, e.g. coronary artery disease (CAD) and myocarditis are leading causes of morbidity and mortality. The prevalence of subclinical heart disease in SLE is unknown. We studied whether a comprehensive cardiovascular magnetic resonance (CMR) protocol may be useful for early diagnosis of heart disease in SLE patients without known CAD

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SLE, as defined by the American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus

Exclusion Criteria:

* age under 18 years
* known coronary artery disease
* impaired renal function with an estimated glomerular filtration rate less than 30 ml/min, estimated by the Modification of Diet in Renal Disease Study Group (MDRD) formula (45)
* devices as pacemakers, implantable cardioverter-defibrillators, insulin pumps and others
* metallic foreign bodies in the eyes, ferromagnetic implants labeled MR unsafe
* allergy against CMR contrast media or adenosine
* presence of chronic atrial fibrillation, 2nd or 3rd degree Atrioventricular (AV)-block, trifascicular block, asthma and severe chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosed SLE
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiovascular pathologies identified by CMR in patients with SLE | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Burkard, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided